CLINICAL TRIAL: NCT05559749
Title: Collaborative Care to Improve Quality of Life for Anxiety and Depression in Epilepsy
Brief Title: Collaborative Care for Anxiety and Depression in Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00088764
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Epilepsy; Anxiety; Depression
Keywords: Quality of Life; Collaborative care
MeSH Terms: conditions — Epilepsy; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-blind hybrid effectiveness-implementation study of a neurology clinic-based 24-week collaborative care intervention versus usual neurology care among a total of 60 adults having epilepsy with anxiety and/or depression symptoms, during 6 months follow-up. Participants will be randomized in a 1:1 ratio to collaborative care intervention versus usual neurology care.
Who Masked: Outcomes Assessor
Masking Description: The randomization table will be prepared by the study statistician, uploaded by the developer, and concealed from the PI and coordinators in the REDCap data management system until after consent, enrollment and baseline data collection is complete, to minimize bias - once participants are randomized it is just outcome assessor who is truly blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- collaborative care (Experimental): The collaborative care team roles include the care manager/social worker and psychiatrist who interact with the patient participant and the patient's neurologist/neurology provider.
  Interventions: Behavioral: collaborative care
- usual neurology care (Active Comparator): Ongoing usual neurology care, without the addition of the collaborative care program - current standard care and is thus an ethically appropriate control condition for effectiveness and implementation trials.
  Interventions: Behavioral: usual neurology care

INTERVENTIONS:
Behavioral: collaborative care — a 24-week neurology based collaborative care program consisting of: 1. a series of every 2 weeks care management calls by the care manager to evaluate anxiety, depression, seizures and side effects and deliver brief therapy interventions to the participant, and 2. collaborative care conferences including a psychiatrist to generate expert recommendations for anxiety and depression management and communication of recommendations between the care manger, psychiatrist and neurologist.
  Arms: collaborative care
Behavioral: usual neurology care — ongoing usual neurology care, without the addition of the collaborative care program
  Arms: usual neurology care

SUMMARY:
This is a randomized effectiveness/implementation trial comparing a 24-week neurology-based collaborative care intervention to usual neurology care among 60 adults with epilepsy.

DETAILED DESCRIPTION:
The intervention is a 24-week, evidence-based collaborative care model initiated around the time of a neurology visit. The collaborative care team roles include the care manager/social worker and psychiatrist who interact with the patient participant and the patient's neurologist/neurology provider.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated Informed Consent Form
* Stated willingness to comply with all study procedures
* Males and Females; Age >= 18 years
* * Diagnosis of epilepsy: Epilepsy diagnosis based on neurology clinician impression or EEG findings
* Anxiety or Depression symptoms
* Receiving clinical neurological care at Atrium Health

Exclusion Criteria:

* Current participation in another treatment of intervention study
* Cognitive limitations precluding completion of Anxiety and Depression self-report instruments on paper, electronically, or by interview
* Comorbid medical condition with life expectancy less than 6 months
* Not a good candidate for collaborative care due to:
* Active ongoing treatment by a psychiatrist
* Active suicidal ideation
* History of past suicide attempt and:
* receiving ongoing psychotherapy OR
* has seen a psychiatrist in the past year
* History of suicide attempt in the past year and:
* currently prescribed 2 or more psychotropic medications for psychiatric indication (not merely as a hypnotic) AND not felt to be a good candidate for collaborative care based on the judgement of the investigators
* Unstable drug or alcohol abuse

For the third Aim (sustainability supplement: intervention only care delivery exploratory study supplement) - the Participants meeting the following criteria may participate

* individuals who meet the above INC-EXC criteria and have completed the Control Arm of a collaborative care research study - NCT05559749 - NCT05353452 or
* individuals who meet the above INC-EXC criteria except rather than having a diagnosis of Epilepsy; they have a diagnosis of functional neurological disorder with seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
change in emotional quality of life subscale of the Quality of Life in Epilepsy Inventory (QOLIE-31) - between two groups | Month 6
  adults with epilepsy and anxiety or depression symptoms - a higher score reflects a more favorable health state

SECONDARY OUTCOMES:
Number of Participants adhering to Intervention | Week 12
  adherence of intervention participants to the majority of care management - proportion of intervention group participants meeting minimum adherence metric of 50% call participation at 12 weeks
Change in Epilepsy-specific quality of life scoring (QOLIE-31) - neurology collaborative care compared to Usual Care | Month 6
  adults with epilepsy and anxiety or depression symptoms - Score ranges from 0-100 with higher score indicating better epilepsy-specific quality of life
Change in the number of depression symptoms - Beck's Depression Inventory (BDI-II) - neurology collaborative care compared to Usual Care | Month 6
  adults with epilepsy and anxiety or depression symptoms -- Depression symptom questionnaire-score ranges from 0-61, with higher score indicating more severe depression symptoms
Change in anxiety symptoms scoring (EASI) Epilepsy Anxiety Survey Instrument - between groups | Month 6
  adults with epilepsy and anxiety or depression symptoms - The score was obtained by computing the sum of the scores obtained by items associated with it, from 0, "not at all", to 3, "nearly every day". The possible total score ranges from 0 to 54, with higher scores indicating worse anxiety symptoms

OTHER OUTCOMES:
Change in Generalized Anxiety Disorders- 7(GAD-7) Score between groups | Month 6
  Questionnaire measuring anxiety symptoms-score ranges from 0 to 21, with higher score indicating increased anxiety symptoms - proportion achieving 50% symptom reduction or remission by 6 months
Change in Neurological Disorders Depression Inventory-Epilepsy (NDDI-E) between groups | Months 3 and 6
  Depression symptom questionnaire specifically for those with epilepsy-score ranges from 6 to 24, with a score >15 indicating presence of a likely major depressive episode.
Change in Patient Health Questionnaire-9 (PHQ-9) Score between groups | Month 6
  Score ranges from 0 to 27, with higher score indicating increased depression symptoms - proportion achieving 50% symptom reduction or remission by 6 months
Emergency Department (ED)/Hospitalization Visits | Month 6
  Number of hospitalizations or visits to ED.
Change in Liverpool Seizure Severity Scale (LSSS) between groups | Month 6
  Seizure severity questionnaire- score ranges from 0 to 100, with higher score indicating increased seizure severity.
Seizure Frequency | Month 6
  Number of seizures experienced by participants - this will be change in seizure frequency and time since last seizure categories from baseline to 6 month follow-up: categorical rating scale developed by Epilepsy Learning Healthcare System & standardized in the American Academy of Neurology (AAN) seizure frequency quality measure
Number of Seizure medication adjustments | Month 6
  number of seizure medication adjustments to address side effects or lack of seizure control over 6 months
Feasibility of Intervention Measure (FIM) Subject Perspective | Baseline and Month 15
  Questionnaire to help determine feasibility of Collaborative Care from Participants' perspectives - score ranges from 5-20, with higher score indication greater feasibility
Feasibility of Intervention Measure (FIM) Neurologist Perspective | Baseline and Month 15
  Questionnaire to help determine feasibility of Collaborative Care from Neurologists' perspectives - score ranges from 5-20, with higher score indication greater feasibility
Acceptability of Intervention Measure (AIM) Subject Perspective | Baseline and Month 15
  Questionnaire to help determine feasibility of Collaborative Care from Participants' perspectives - score ranges from 5-20, with higher score indication greater acceptability
Acceptability of Intervention Measure (AIM) Neurologist Perspective | Baseline and Month 15
  Questionnaire to help determine feasibility of Collaborative Care from Neurologists' perspectives - score ranges from 5-20, with higher score indication greater acceptability
Intervention Appropriateness Measure (IAM) Subject Perspective | Baseline and Month 15
  Questionnaire to help determine appropriateness of Collaborative Care from participants' perspectives. Score ranges form 5-20 with higher score indication greater appropriateness
Intervention Appropriateness Measure (IAM) Neurologist Perspective | Baseline and Month 15
  Questionnaire to help determine appropriateness of Collaborative Care from Neurologists' perspectives. Score ranges form 5-20 with higher score indication greater appropriateness
Individual Participant Collaborative Care Call Attendance Percentage | Weeks 12 and 24
  Individual Participant Collaborative Care Call Attendance Percentage
change in emotional quality of life subscale of the Quality of Life in Epilepsy Inventory (QOLIE-31) - between two groups | Month 3
  adults with epilepsy and anxiety or depression symptoms - a higher score reflects a more favorable health state
change in brEASI (Brief anxiety in epilepsy survey instrument) | Months 3 and 6
  Scores of ≥7 on the Brief anxiety in epilepsy survey instrument (brEASI) indicate probable anxiety disorder. Scores range from 0 to 24, with higher scores indicting increased anxiety symptoms.
Beck Depression Inventory (BDI) change | Month 6
  proportion achieving 50% symptom reduction or remission by 6 months
anxiety in epilepsy survey instrument (EASI) change | Month 6
  proportion achieving 50% symptom reduction or remission by 6 months
Sustainability - insurance payment (quantity) for collaborative care billing codes | Month 6
  only measured in Aim 3 - sustainability supplement - intervention only clinical care delivery with insurance billing
Sustainability - did insurance pay (yes/no) for collaborative care billing | Month 6
  only measured in Aim 3 - sustainability supplement - intervention only clinical care delivery with insurance billing

CONTACTS AND LOCATIONS:
Overall Officials: Heidi M Munger Clary, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and results published by primary study team, de-identified, archived data will be stored for potential use if requested by other qualified researchers including those outside of the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after results published by primary study team
Access Criteria: Access to study data may be provided by the PI if requested by qualified investigators for individual participant data meta-analyses or potentially for other methodologically sound proposals.